CLINICAL TRIAL: NCT02685748
Title: Aspirin as Adjuvant Therapy in Young Psychotic Patients
Brief Title: Aspirin in Young Psychotic Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Clinic for Psychiatric Disorders, Dr Laza Lazarevic (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dragana Pavićević, Dr Dragana Pavicevic, Clinic for Psychiatric Disorders, Dr Laza Lazarevic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #15T-006
Record Dates: First submitted 2016-02-08; First posted 2016-02-19 (Estimated); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Psychosis; Acute Psychosis; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Aspirin; Sugars; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin & pantoprazole (Experimental): Aspirin 1000 mg/pd per os in two doses
  Pantoprazole 40 mg/pd per os in two doses for gastric protection
  Interventions: Drug: Aspirin; Drug: Pantoprazole
- Placebo (Placebo Comparator): Two pills in the morning and two in the evening
  All pills (aspirin, pantoprazole an placebo) will be the same looking- in the same capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 1000 mg pd in two doses
  Other Names: Acetylsalicylic acid
  Arms: Aspirin & pantoprazole
Drug: Placebo — two pills twice a day (instead of aspirin and pantoprazole)
  Other Names: sugar pill
  Arms: Placebo
Drug: Pantoprazole — Pantoprazole 40 mg/pd in two doses, for gastric protection
  Other Names: Protonix; Controloc
  Arms: Aspirin & pantoprazole

SUMMARY:
In this double blind randomized clinical trial the investigators are going to exam influence of adjuvant Aspirin therapy on soft neurological signs (Heidelberg scale), positive and negative symptoms (PANSS), cytokine profile and inflammatory factors, as well as on cognition (MoCA) in young psychotic patients.

DETAILED DESCRIPTION:
Schizophrenia as psychiatric paradigm is one of the most mysterious mental illness, for decades remains a challenge to many clinicians and researchers with its complex, fundamental mechanisms.

Soft neurological signs (SNS) are described as non-localized neurological abnormalities that cannot be associated with damage of a specific brain region. It is believed that they are not part of a well-defined neurological syndrome. They include neurological abnormalities with deficits in sensory integration, motor coordination and sequencing of complex motor acts. They have a higher prevalence in schizophrenic patients compared to healthy population. Moreover, SNS have been consistently demonstrated in neuroleptic naive patients in the first episode of illness. There is also an increased prevalence in non- schizophrenic relatives of patients with schizophrenia. It is considered that they are not potentiated by antipsychotics. For all these reasons it is believed that they are the inherent quality of schizophrenia - "trait" marker, or endophenotypes.

According to the so-called "Two hit" hypothesis in the development of schizophrenia, there are two periods of increased vulnerability. The first one is in a fetal age when it comes to the interaction of genetic and environmental factors such as infection and inflammatory processes who may also serve this function. The second period of vulnerability is a period of adolescence, or early adult age when the influence of environmental factors leads to clinical manifestations of the disease. It is thought that cytokines have key role in the first strike.

Cytokines are mediators of communication between the neural elements in all aspects of the development of the nervous system. Until now, numerous studies indicated modification of specific cytokines in psychotic disorders and their possible role in the proposed concept of "microglial hypothesis" of schizophrenia. Hypothesis of activation Th1 and Th2 immune response, with a predominance of Th2 immune response is proposed in schizophrenia. Type-17 cytokines are important in mediating tissue damage in autoimmune diseases. Regulatory cytokines suppress immune responses and maintain self-tolerance.

Consequently, the question is whether the combination of antipsychotic drugs with anti-inflammatory drugs is more useful than independent antipsychotic therapy? Laan and colleagues in 2010. carried out a randomized, double- blind, placebo - controlled study to determine if the adjuvant aspirin therapy could be useful for patients who are already taking antipsychotics. They concluded that the therapy antipsychotic + aspirin was significantly superior to placebo + antipsychotic therapy. PANSS score was significantly lower in the aspirin group.

The aim of the study would be to determine the effects of adjuvant aspirin therapy on Soft Neurological Signs, PANSS and the cytokine profile. The investigators expect the reduction of PANSS scores in both groups of patients (aspirin group and placebo group). If there is no significant changes of SNS between groups, the results would support SNS as trait characteristics of schizophrenia.

The research would be done on hospitalized patients at the Clinic for Psychiatric Disorders "Dr Laza Lazarevic" in Belgrade. Part of the study (immunology) will be done on Medical Faculty University of Kragujevac.

The study would be a randomized, double-blind, placebo controlled in two parallel groups of 50 to 60 patients who are neuroleptic naive or previously minimally medicated (in the past 6 months without any antipsychotic treatment) with the duration of the illness up to seven years. The study would involve the patients of both sexes, aged 18 to 28 years, according to ICD 10 (10th revision of the International Statistical Classification of Diseases and Related Health Problems) criteria to satisfy diagnosis F 20 to F 29. Each patient who enters the hospital and meets the inclusion criteria would be taken into consideration. If patient satisfies exclusion criteria and sign consent, then s/he would be randomized into two groups: Experimental group (antipsychotic + aspirin) and Control group (antipsychotic + placebo). Patients in experimental group (EG) would receive 1,000 mg of aspirin pro die and pantoprazole 40 mg pro die in two doses for gastric protection.

Only one researcher would know in which group patient belongs (would be responsible only for randomization, would not be rater or treating psychiatrist). The same researcher would give boxes with medications marked with the patient's name. In fact, all medications (aspirin, pantoprazole, and placebo) would be packaged in the same looking capsules.

The protocol would consist of three planned visits for patients in both groups. On the first visit blood samples would be taken for the implementation of immunological tests as well as for laboratory inflammatory factors; patients would be subjected to clinical psychiatric and physical examination, BMI measurement; PANSS scale will be done. After calming the signs of acute psychosis, on 3rd day, patients would be examined with Heidelberg and MoCA scale; patients would start to take Aspirin or Placebo. At the end of 6th week from the second visit (+/- 3 days), on the third visit, blood samples would be taken again for analyzing cytokine profile and inflammatory factors. PANSS, Heidelberg and MoCA scales would be performed again.

The investigators would consider the following factors: patient sex, age of the patients, clinical characteristics, the role of heredity, type of therapy/ prescribed typical or atypical antipsychotic; side effects of treatment and type of treatment response. Serum concentrations of cytokines will be examined with commercial ELISA tests.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 28 years of life
* diagnostic categories from F 20 to F 29, according to ICD 10 (International Classification of Diseases Version 10) criteria
* duration of illness ≤ 7 years

Exclusion Criteria:

* Substance abuse
* Primary cognitive impairment
* Contraindications and special caution for acetylsalicylic acid and pantoprazole: hypersensitivity to aspirin and other NSAIDs or pantoprazole, ulcers, gastritis, pregnancy, haemophilia, bleeding disorders, gout, asthma, COPD (Chronic obstructive pulmonary disease), bronchospasm induced by NSAIDs, angioedema, urticaria, haemolytic anaemia, use of warfarin or methotrexate, diabetes, reduced function of liver and/or kidney, heart failure, surgical/dental intervention, interactions with certain psychotropic drugs

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragana Pavićević, psychiatrist, Principal Investigator — Clinic for psychiatric disorder Dr Laza Lazarević
Locations (1):
- Clinic for psychiatric disorders Dr Laza Lazarevic, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results of study:
  * scores of PANSS (cumulative positive, negative and general scores)
  * MoCA scale cumulative scores
  * Heidelberg scale cumulative scores
  * as well as levels of CRP, WBC and cytokines.
Supporting Information: Study Protocol, SAP
Time Frame: Starting in January 2024. for 24 months.
Access Criteria: Investigators who proposed use of data has been approved by an independent review committee for meta analysis.

REFERENCES:
- [Background] Mayoral M, Bombin I, Castro-Fornieles J, Gonzalez-Pinto A, Otero S, Parellada M, Moreno D, Baeza I, Graell M, Rapado M, Arango C. Longitudinal study of neurological soft signs in first-episode early-onset psychosis. J Child Psychol Psychiatry. 2012 Mar;53(3):323-31. doi: 10.1111/j.1469-7610.2011.02475.x. Epub 2011 Oct 25. PMID 22023091
- [Background] Bombin I, Arango C, Buchanan RW. Significance and meaning of neurological signs in schizophrenia: two decades later. Schizophr Bull. 2005 Oct;31(4):962-77. doi: 10.1093/schbul/sbi028. Epub 2005 Jun 15. PMID 15958818
- [Background] Heinrichs DW, Buchanan RW. Significance and meaning of neurological signs in schizophrenia. Am J Psychiatry. 1988 Jan;145(1):11-8. doi: 10.1176/ajp.145.1.11. PMID 3276226
- [Background] Hirjak D, Wolf RC, Koch SC, Mehl L, Kelbel JK, Kubera KM, Traeger T, Fuchs T, Thomann PA. Neurological abnormalities in recent-onset schizophrenia and asperger-syndrome. Front Psychiatry. 2014 Aug 6;5:91. doi: 10.3389/fpsyt.2014.00091. eCollection 2014. PMID 25147527
- [Background] Schroder J, Niethammer R, Geider FJ, Reitz C, Binkert M, Jauss M, Sauer H. Neurological soft signs in schizophrenia. Schizophr Res. 1991 Dec;6(1):25-30. doi: 10.1016/0920-9964(91)90017-l. PMID 1786233
- [Background] Bachmann S, Bottmer C, Schroder J. Neurological soft signs in first-episode schizophrenia: a follow-up study. Am J Psychiatry. 2005 Dec;162(12):2337-43. doi: 10.1176/appi.ajp.162.12.2337. PMID 16330599
- [Background] Maynard TM, Sikich L, Lieberman JA, LaMantia AS. Neural development, cell-cell signaling, and the "two-hit" hypothesis of schizophrenia. Schizophr Bull. 2001;27(3):457-76. doi: 10.1093/oxfordjournals.schbul.a006887. PMID 11596847
- [Background] Feigenson KA, Kusnecov AW, Silverstein SM. Inflammation and the two-hit hypothesis of schizophrenia. Neurosci Biobehav Rev. 2014 Jan;38:72-93. doi: 10.1016/j.neubiorev.2013.11.006. Epub 2013 Nov 15. PMID 24247023
- [Background] Mousa A, Bakhiet M. Role of cytokine signaling during nervous system development. Int J Mol Sci. 2013 Jul 4;14(7):13931-57. doi: 10.3390/ijms140713931. PMID 23880850
- [Background] Monji A, Kato T, Kanba S. Cytokines and schizophrenia: Microglia hypothesis of schizophrenia. Psychiatry Clin Neurosci. 2009 Jun;63(3):257-65. doi: 10.1111/j.1440-1819.2009.01945.x. PMID 19579286
- [Background] Avgustin B, Wraber B, Tavcar R. Increased Th1 and Th2 immune reactivity with relative Th2 dominance in patients with acute exacerbation of schizophrenia. Croat Med J. 2005 Apr;46(2):268-74. PMID 15849849
- [Background] Borovcanin M, Jovanovic I, Radosavljevic G, Djukic Dejanovic S, Bankovic D, Arsenijevic N, Lukic ML. Elevated serum level of type-2 cytokine and low IL-17 in first episode psychosis and schizophrenia in relapse. J Psychiatr Res. 2012 Nov;46(11):1421-6. doi: 10.1016/j.jpsychires.2012.08.016. Epub 2012 Sep 10. PMID 22974591
- [Background] Borovcanin M, Jovanovic I, Radosavljevic G, Djukic Dejanovic S, Stefanovic V, Arsenijevic N, Lukic ML. Antipsychotics can modulate the cytokine profile in schizophrenia: attenuation of the type-2 inflammatory response. Schizophr Res. 2013 Jun;147(1):103-109. doi: 10.1016/j.schres.2013.03.027. Epub 2013 Apr 16. PMID 23602340
- [Background] Laan W, Grobbee DE, Selten JP, Heijnen CJ, Kahn RS, Burger H. Adjuvant aspirin therapy reduces symptoms of schizophrenia spectrum disorders: results from a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2010 May;71(5):520-7. doi: 10.4088/JCP.09m05117yel. PMID 20492850
- [Background] Sommer IE, van Westrhenen R, Begemann MJ, de Witte LD, Leucht S, Kahn RS. Efficacy of anti-inflammatory agents to improve symptoms in patients with schizophrenia: an update. Schizophr Bull. 2014 Jan;40(1):181-91. doi: 10.1093/schbul/sbt139. Epub 2013 Oct 8. PMID 24106335
- See also: Stoyanova M, Hranov L. Soft neurological signs in patients with bipolar disorder. European Psychiatry, 2014: 29 (1) 1 — http://dx.doi.org/10.1016/S0924-9338(14)78043-5
- See also: Schröder J, Heuser M. Neurological Soft Signs in First -Episode Schizophrenia. Directions in Psychiatry 2008, Vol. 28 (19): 243-57. — https://www.klinikum.uni-heidelberg.de/fileadmin/gerontopsychiatrie/pdf/2008_Schroeder_Neurol_soft_signs_in_first-episode_schizophrenia.pdf
- See also: Howard, J. (2013) The cytokine hypothesis: A neurodevelopmental explanation for the emergence of schizophrenia later in life. Advances in Bioscience and Biotechnology, 4, 81-88 — http://file.scirp.org/Html/11-7300647_36227.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 patients enrolled, 57 randomized
Groups:
- Aspirin: Aspirin 1000 mg/per day, orally, two doses
  Pantoprazole 40 mg/per day, orally, in two doses for gastric protection
- Placebo: placebo- two times a day two pills orally
Period: Overall Study
Arm/Group | Aspirin | Placebo
Started | 28 | 29
Completed | 25 | 27
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Aspirin: Aspirin 1000 mg/pd per os in two doses
  Pantoprazole 40 mg/pd per os in two doses for gastric protection
- Placebo: placebo- 2 times a day two pills
- Total: Total of all reporting groups
Arm/Group | Aspirin | Placebo | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 29 | 57
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 29 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 29 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Neurological Soft Signs
Description: Neurological soft signs were assessed with the Heidelberg Scale which consists of five subscales (motor coordination, integrative functions, complex motor tasks, orientation, hard signs) comprising 16 items (gait, tandem walking, right/left orientation, arm holding test, finger to nose test, Ozeretzki's test, diadochokinesis, pronation-supination, finger to thumb opposition, mirror movements, two point discrimination, graphaesthesia, face- hand test, stereognosis, fist- edge- palm test, speech and articulation).
  Ratings are given on a 0-3 point scale (no/slight/moderate/marked abnormality, respectively) for all items except for tandem walking (0-1 point scale; 0: no/slight, 1: moderate/marked abnormality). Scale ranges: minimum- 0 (better outcome), maximum 46 points (worse outcome).
Time Frame: Comparison of total scores on Heidelberg scale between groups (aspirin and placebo group) after 6 weeks of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aspirin: Aspirin 1000 mg/ per day, orally, in two doses
  Pantoprazole 40 mg/ per day, orally, in two doses for gastric protection
  Aspirin: 1000 mg/ per day, orally, in two doses
  Pantoprazole: Pantoprazole 40 mg/ per day, orally, in two doses, for gastric protection
- Placebo: Two pills in the morning and two in the evening
  All pills (aspirin, pantoprazole an placebo) will be the same looking- in the same capsules.
  Placebo: two pills twice a day (instead of aspirin and pantoprazole)
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 25 | 27
score on a scale | 6.96 (1.670) | 7.04 (1.537)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Other; p = 0.863, t-test, 2 sided; Mean Difference (Final Values) = -0.077, 95% CI 2-sided [-0.969 to 0.815], Standard Error of Mean 0.444

2. Primary Outcome: Psychopathology Symptoms Assessed by PANSS
Description: The Positive and Negative Syndrome Scale (PANSS) is 30 item scale used to evaluate the presence, absence and severity of Positive, Negative and General Psychopathology symptoms of schizophrenia. Ratings are given on a 1-7 point scale (1- absent, 2- minimal, 3- mild, 4- moderate, 5- moderate severe, 6- severe, 7- extreme). Patient can not score lower than 30 for the total PANSS score. Maximum score is 210.
  Higher scores mean a worse outcome.
Time Frame: Comparison of total scores on PANSS (aspirin and placebo group) after 6 weeks of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Aspirin: Aspirin: 1000 mg pd in two doses
  Pantoprazole: Pantoprazole 40 mg/pd in two doses, for gastric protection
- Placebo: Two pills in the morning and two in the evening
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 25 | 27
score on a scale | 67.70 (10.227) | 71.32 (6.549)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Other — T test for independent samples; p = 0.133, t-test, 2 sided; Mean Difference (Final Values) = 3.616, 95% CI 2-sided [-1.147 to 8.379], Standard Error of Mean 2.364

3. Secondary Outcome: Cognitive Assessment by MoCA Scale
Description: The Montreal Cognitive Assessment (MoCA) is a test used to detect cognitive decline. The MoCA test examines seven domains (executive/visuospatial function, naming, attention, language, abstraction, recall, and orientation) of cognitive function with a total of 11 questions with a maximum score of 30. A score of 26 or over is considered to be normal. A score of less than 26 indicates cognitive impairment (worse outcome). Minimal score is 0.
Time Frame: Comparison of total scores on MoCA scale (aspirin and placebo group) after 6 weeks of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 25 | 27
score on a scale | 27.63 (1.282) | 28.32 (1.757)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Other; p = 1.607, t-test, 2 sided; Mean Difference (Final Values) = 0.114, 95% CI 2-sided [-1.1553 to 0.172], Standard Error of Mean 0.430

4. Secondary Outcome: Marker of Inflammation: C-reactive Protein (CRP)
Description: A C-reactive protein (CRP) test measures the level of C-reactive protein - a protein made by liver and releases in bloodstream in response to inflammation. Levels below 5 milligrams per liter (mg/L) are usually considered normal or free from infections.
Time Frame: Comparison of CRP levels between groups (aspirin and placebo group) after six weeks of treatment.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 25 | 27
mg/L | 3.080 (2.5549) | 4.363 (8.417)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Other; p = 0.468, t-test, 2 sided; Mean Difference (Final Values) = -1.282, 95% CI 2-sided [-4.807 to 2.241], Standard Error of Mean 1.754

5. Secondary Outcome: Marker of Inflammation- White Blood Cells (WBC)
Description: A white blood cell (WBC) count is a test that measures the number of white blood cells in blood. A white blood cell count can detect infections within body. The normal white blood cell count ranges between 4,000 and 11,000 cells per microliter.
Time Frame: Comparison of WBC levels (aspirin and placebo group) after 6 weeks of treatment.
Measure: Mean (Standard Deviation); unit: x 1000 cells per microliter
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 25 | 27
x 1000 cells per microliter | 6.252 (1.528) | 6.303 (1.405)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Other; p = 0.899, t-test, 2 sided; Mean Difference (Final Values) = -0.051, 95% CI 2-sided [-0.869 to 0.765], Standard Error of Mean 0.406

6. Secondary Outcome: Cytokine Profile- Th1- Interferon Gamma (IFN-γ)
Description: Change of Interferon Gamma (IFN-γ) immune response
Time Frame: Comparison of IFN Gamma levels (aspirin and placebo group) after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: pg/l
Groups:
- Placebo: Placebo: two pills twice a day
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 25 | 27
pg/l | 92.557 (29.696) | 85.507 (18.420)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Other; p = 0.305, t-test, 2 sided; Mean Difference (Final Values) = 7.050, 95% CI 2-sided [-6.602 to 20.703], Standard Deviation 6.797

7. Secondary Outcome: Cytokine Profile- Th2-Interleukin 4 (IL4)
Description: Change of IL4 immune response
Time Frame: Comparison of IL 4 levels (aspirin and placebo group) after 6 weeks of treatment
Population: patients who have completed study
Measure: Mean (Standard Deviation); unit: pg/l
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 25 | 27
pg/l | 620.340 (817.873) | 460.042 (133.44)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Other; p = 0.320, t-test, 2 sided; Mean Difference (Final Values) = 160.298, 95% CI 2-sided [-160.118 to 480.714], Standard Error of Mean 159.525

8. Secondary Outcome: Cytokine Profile- Type 17- Interleukin 17 (IL17)
Description: Change of IL17 immune response
Time Frame: Comparison of IL 17 levels (aspirin and placebo group) after 6 weeks of treatment
Population: patients who have completed study
Measure: Mean (Standard Deviation); unit: pg/l
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 25 | 27
pg/l | 11.760 (14.691) | 13.255 (10.809)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; Test type: Other; p = 0.676, t-test, 2 sided; Mean Difference (Final Values) = -1.495, 95% CI 2-sided [-8.642 to 5.651], Standard Error of Mean 3.558

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Aspirin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

LIMITATIONS AND CAVEATS:
Acute phase of disorder, small number of patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT02685748/Prot_SAP_ICF_001.pdf